CLINICAL TRIAL: NCT06468852
Title: Effect of Goal-Directed Fluid Therapy on the Postoperative Outcome in Head and Neck Cancer Surgery: A Randomized Controlled Trial
Brief Title: GDFT on the Postoperative Outcome in Head and Neck Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TREC2024-KY059
Record Dates: First submitted 2024-06-04; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Complications
Keywords: Postoperative Complications; Early Goal-Directed Therapy; Fluid therapy; Head and Neck Neoplasms
MeSH Terms: conditions — Postoperative Complications; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients were unaware of their group allocation. Due to the presence of the cardiac index trend monitoring device, care providers who supported to fluid strategy administration in the operating room could not be blinded. The outcomes assessor were blinded to the allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDFT group (Experimental): Patients in GDFT group will receive GDFT protocol, Stroke volume variation (SVV)≤12% and cardiac index (CI)≥2.5L/min/m2 are the goals of fluid therapy, while the mean arterial pressure (MAP) are kept between 65 and 90 mmHg. 5mL/kg of crystalloids will be infused during induction period, followed by an infusion rate of 2 mL/kg/h to supplement the physiological requirements. If SVV>12% for more than 5 min, a 250 mL bolus of colloid is given. Another 250 ml bolus of colloid is administrated if SVV was still more than 12% or SV decreased over 10%. If the CI<2.5 L/min/m2, inotropes are used to achieve this minimum CI, serving as a safety parameter to prevent the patient from being exposure to a low cardiac output state. If SVV and CI reached the s target range but MAP could not maintain the expected level, vasopressors were started. Assess the patients every 5min intraoperatively to ensure that all parameters adhere to the target range according to the study algorithm.
  Interventions: Procedure: Goal-Directed Fluid Therapy
- conventional fluid therapy group (No Intervention): Patients in conventional fluid therapy group, fluid management will be carried out according to the clinical practice routine, maintaining MAP≥65mmHg and urine output ≥0.5ml/kg/h, intraoperatively. When the anesthesiologist empirically determines that the fluid infusion is sufficient but MAP does not maintain the expected level, vasopressor or inotropic drugs are given to maintain the blood pressure.

INTERVENTIONS:
Procedure: Goal-Directed Fluid Therapy — Stroke volume variation (SVV)≤12% and cardiac index (CI)≥2.5L/min/m2 are the goals of Goal-Directed fluid therapy, while the mean arterial pressure (MAP) are kept between 65 and 90 mmHg. 5mL/kg of crystalloids will be infused during induction period, followed by an infusion rate of 2 mL/kg/h to supplement the physiological requirements. If SVV>12% for more than 5 min, a 250 mL bolus of colloid is given. Another 250 ml bolus of colloid is administrated if SVV was still more than 12% or SV decreased over 10%. If the CI<2.5 L/min/m2, inotropes are used to achieve this minimum CI, serving as a safety parameter to prevent the patient from being exposure to a low cardiac output state. If SVV and CI reached the s target range but MAP could not maintain the expected level, vasopressors were started. Assess the patients every 5min intraoperatively to ensure that all parameters adhere to the target range according to the study algorithm.
  Arms: GDFT group

SUMMARY:
The goal of this clinical trial is to evaluate whether goal-directed fluid therapy (GDFT) can improve the postoperative recovery in patients undergoing head and neck cancer surgery. It aims to answer is:

• Whether GDFT can reduce the occurrence of serious postoperative complications? Researchers will compare GDFT protocol to a standard conventional fluid therapy in head and neck cancer surgery to see if GDFT strategy works to improve the postoperative recovery.

Participants will

* Receive GDFT protocol or a conventional fluid therapy during the surgery.
* Be continuously follow-up during hospitalization and after discharge to record the occurrence of postoperative complications.

DETAILED DESCRIPTION:
Postoperative complications have become the main cause of prolonged hospitalization and reduced postoperative survival rate among surgical patients. Goal-Directed Fluid Therapy (GDFT) has been reported to reduce the incidence of postoperative complications and mortality, shorten the hospital stay, and improve the outcome in major abdominal surgery patients. However, the benefit of the GDFT in patients undergoing head and neck surgery remains controversial. The purpose of this study is to evaluate whether GDFT can reduce the occurrence of serious postoperative complications and shorten the postoperative hospital stay, compared with a standard conventional fluid therapy in patients undergoing head and neck cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (Age≥18)
* Scheduled to undergo head and neck cancer surgery (including nasopharyngeal carcinoma, laryngocarcinoma, hypopharyngeal carcinoma, and other head and neck malignancies, but not thyroid cancer) with an expected duration of 2 hours or longer
* Agree to receive invasive artery blood pressure monitoring

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) classification>Ⅳ
* Palliative surgery was performed for the terminal tumors
* Microlaryngoscopic laser surgery or endoscopic surgery
* Underwent major thoracic or abdominal surgery within 30 days
* Regular renal replacement therapy is required
* NYHA grade>3 or ejection fraction <30%
* Lung disease does not tolerate the tidal volume by 8 ml/kg
* Atrial fibrillation
* Unable to give informed consent
* pregnant or lactating woman
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Serious complications occurred within 30 days after surgery | within 30 days after surgery
  Unit: %; All postoperative complications will be evaluated according the Clavien-Dino classification(CDc) of surgical complications. Each complication has an equal weight, and patients with at least one complication will be considered to have experienced postoperative complications.
  The serious postoperative complications were defined as CDc≥3.

SECONDARY OUTCOMES:
All complications within 30 days after surgery | within 30 days after surgery
  Unit: %;All postoperative complications will be evaluated according the Clavien-Dino classification(CDc) of surgical complications.
The length of hospital stay after surgery | 1 months after operation
  Unit: days; from date of operation till date of discharge
Cost of hospitalization | 1 months after operation
  Unit: yuan; Total cost during hospitalization
Quality of Recovery Score | At 1,3, and 5 days after surgery
  Unit: point; Use QoR-15 to evaluate the postoperative recovery of all patients. QoR-15 is a global measure of recovery after surgery that evaluates five dimensions of recovery: physical comfort (5 items), physical independence (2 items), emotional state (4 items), psychological support (2 items), and pain (2 items). Each item is rated on an 11- point scale based on its frequency on the questionnaire (greater score at greater frequency for positive items and less frequency for negative items). The total score ranged from 0 (poorest recovery quality) to 150 (best recovery quality).

CONTACTS AND LOCATIONS:
Overall Officials: Guyan Wang, Principal Investigator — Beijing Tongren Hospital, CMU
Locations (1):
- Beijing tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] McMahon JD, MacIver C, Smith M, Stathopoulos P, Wales C, McNulty R, Handley TP, Devine JC. Postoperative complications after major head and neck surgery with free flap repair--prevalence, patterns, and determinants: a prospective cohort study. Br J Oral Maxillofac Surg. 2013 Dec;51(8):689-95. doi: 10.1016/j.bjoms.2013.04.015. Epub 2013 May 31. PMID 23727043
- [Background] Loeffelbein DJ, Julinek A, Wolff KD, Kochs E, Haller B, Haseneder R. Perioperative risk factors for postoperative pulmonary complications after major oral and maxillofacial surgery with microvascular reconstruction: A retrospective analysis of 648 cases. J Craniomaxillofac Surg. 2016 Aug;44(8):952-7. doi: 10.1016/j.jcms.2016.05.007. Epub 2016 May 14. PMID 27259678
- [Background] Liang X, Chen X, Wang G, Wang Y, Shi D, Zhao M, Zheng H, Cui X. Intraoperative hypotension, oliguria and operation time are associated with pulmonary embolism after radical resection of head and neck cancers: a case control study. BMC Anesthesiol. 2021 Dec 3;21(1):304. doi: 10.1186/s12871-021-01521-4. PMID 34856931
- [Background] Dushianthan A, Knight M, Russell P, Grocott MP. Goal-directed haemodynamic therapy (GDHT) in surgical patients: systematic review and meta-analysis of the impact of GDHT on post-operative pulmonary complications. Perioper Med (Lond). 2020 Oct 15;9:30. doi: 10.1186/s13741-020-00161-5. eCollection 2020. PMID 33072306
- [Background] Sun Y, Chai F, Pan C, Romeiser JL, Gan TJ. Effect of perioperative goal-directed hemodynamic therapy on postoperative recovery following major abdominal surgery-a systematic review and meta-analysis of randomized controlled trials. Crit Care. 2017 Jun 12;21(1):141. doi: 10.1186/s13054-017-1728-8. PMID 28602158
- [Background] Reiterer C, Kabon B, Zotti O, Obradovic M, Kurz A, Fleischmann E. Effect of goal-directed crystalloid- versus colloid-based fluid strategy on tissue oxygen tension: a randomised controlled trial. Br J Anaesth. 2019 Dec;123(6):768-776. doi: 10.1016/j.bja.2019.08.027. Epub 2019 Oct 15. PMID 31627889
- [Derived] Liang X, Xi C, Zhou H, Wang S, Shi D, Wang Y, Shen W, Wang G. Effect of goal-directed fluid therapy on the postoperative outcome in head and neck cancer surgery: study protocol for a randomized controlled trial. Trials. 2025 Oct 15;26(1):412. doi: 10.1186/s13063-025-09152-7. PMID 41094585

DOCUMENTS (1):
  • Informed Consent Form (2024-05-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT06468852/ICF_000.pdf